CLINICAL TRIAL: NCT04074408
Title: Intracavitary Injection of Human Umbilical Cord Mesenchymal Stem Cells in Acute Basal Ganglia Hematoma After Stereotactic Aspiration: a Randomized, Single-blind, Placebo-Controlled, Phase 2 Trial
Brief Title: Intracavitary Injection of hUMSCs in Acute Basal Ganglia Hematoma After Stereotactic Aspiration
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital, University of Science and Technology of China (Other); Zhejiang University (Other); First Affiliated Hospital of Fujian Medical University (Other); Jinhua Hospital, School of Medicine, Zhejiang University (Unknown); Taizhou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZJU-hUMSCs
Record Dates: First submitted 2019-08-26; First posted 2019-08-30 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2019-08

CONDITIONS: Basal Ganglia Hematoma
MeSH Terms: conditions — Basal Ganglia Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Masking Description: The hUMSCs suspension and placebo solvent have different appearance so only the participants but not the researches can be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): low dose hUMSCs or high dose hUMSCs
  Interventions: Procedure: stereotactic surgery; Biological: hUMSCs
- Cohort 2 (Experimental): best dose of hUMSCs (from cohort 1) or placebo
  Interventions: Procedure: stereotactic surgery; Biological: hUMSCs; Biological: placebo

INTERVENTIONS:
Procedure: stereotactic surgery — stereotactic aspiration surgery
Biological: hUMSCs — single intracavitary infusion 1 day after stereotactic aspiration surgery
Biological: placebo — single intracavitary infusion 1 day after stereotactic aspiration surgery
  Arms: Cohort 2

SUMMARY:
A study to examine the safety and potential effectiveness of human umbilical cord mesenchymal stem cells (hUMSCs) in adults who have suffered spontaneous cerebral hemorrhage in basal ganglia. The hypothesis is that hUMSCs will be safe and can improve neurological function after intracerebral hemorrhage so that improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 30 and 75 years of age, diagnosed of spontaneous basal ganglia hemorrhage by imaging (CT, CTA, etc.) with a volume from 10 ml to 60 ml calculated by ABC/2 formula.
* Within 5 days from onset to operation, and no improvement.
* Glasgow Coma Scale (GCS) score of 9 to 15.
* With dysfunction such as hematoma-related motor aphasia, sensory aphasia, hemiplegic limb muscle strength≤grade 3.
* Modified Rankin scale (mRS) score≤1 in past medical history.
* Women of reproductive age have negative pregnancy tests.
* The participants or the legal guardian/representative who are suitable and willing to participate in the clinical trial and can cooperate to complete the follow-ups.

Exclusion Criteria:

* Imaging-based diagnosis of cerebrovascular abnormalities such as ruptured aneurysm, arteriovenous malformation AVM and moyamoya disease as well as hemorrhagic transformation of ischemic infarct and recent recurrence (within 1 year) of cerebral hemorrhage.
* In the sequela stage of cerebral trauma.
* Hematoma involves other structures including but not limited to the thalamus and midbrain or complicated with intraventricular hemorrhage.
* With neurologic impairment before cerebral hemorrhage onset.
* Participants receiving anticoagulant or antiplatelet therapy.
* The disease progresses quickly. Manifestation of cerebral herniation such as bilateral dilated pupil, disappearance of light reflex, and unstable vital signs.
* Active stage of infectious diseases including but not limited to HIV, hepatitis B, and C.
* History of poorly controlled seizures.
* History of severe co-morbidity (including but not limited to hepatic, renal, gastrointestinal, respiratory, cardiovascular, endocrine, immune and/or hematological disorders) which may affect the outcome assessment. Coagulation dysfunction INR >1.4, PTT>37 seconds, thrombocytopenia (PLT<8×10^9/L), serum creatinine exceeded the upper limit of normal by 1.4 times, serum ALT >150U/L, and/or serum total bilirubin >1.6mg/dl.
* Participants with a mechanical heart valve. Biological valves are acceptable.
* Participants with a risk of embolism (including but not limited to a history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis or subacute bacterial endocarditis). Atrial fibrillation without mitral stenosis is acceptable.
* May be pregnant in the near future or already pregnant.
* Enrolled in this clinical trial or participating in other interventional medical research or clinical trials at the same time.
* Participants difficult to follow up or with poor compliance due to various reasons (including but not limited to geographical and social factors, drug or alcohol abuse).
* Participants or the legal guardian/representative is unable or unwilling to give the written informed consent.
* Vulnerable groups (including but not limited to mental retardation, abuse, inability to fully exercise informed consent).
* Any subject that the researchers think is not suitable for enrollment.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose limiting adverse events | 3 days
Modified Rankin Scale (mRS) to measure the prognosis | 3 months
  The Modified Rankin Scale (mRS) measures independence rather than performance of specific tasks. Scale consists of six grades from 0 to 5; 0 denotes no symptoms and 5 indicates severe disability. For clinical purpose, mild disability range is from 0 to 2; moderate disability ranges from 3 to 4 and 5 indicates severe disability.
National institute of Health Stroke Scale (NIHSS) to measure stroke recovery | 3 months
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item impairment scale used to measure stroke severity. The NIHSS includes the following domains: level of consciousness, eye movements, integrity of visual fields, facial movements, arm and leg muscle strength, sensation, coordination, language, speech and neglect. Each impairment is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke).
Barthel Index (BI) to evaluate the self-care ability | 3 months
  The Barthel index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). It uses ten variables describing ADL and mobility including: help needed with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, bathing, presence of absence of fecal incontinence and urinary incontinence. Each performance item is rated on this scale with a given number of points from 0 to 10 or 0 to 15. Item scores are summed to a total score ranging from 0 to 100. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence. Totally dependent ranges from 0 to 20, severe dependent ranges from 21 to 60, moderate dependent ranges from 61 to 90, mild dependent ranges from 91 to 99, and 100 indicates completely independent.
Rate of muscle strength level of the hemiplegic limb | 3 months

SECONDARY OUTCOMES:
Mortality rate | 12 months
Change in Glasgow coma scale (GCS) score | 1 month
  The Glasgow coma scale (GCS) is based on a 15-point scale for estimating and categorizing the consciousness. The test measures the motor response (1 to 6), verbal response (1 to 5) and eye opening response (1 to 4). The score is determined by the sum of the score in each of the 3 categories, with a maximum score of 15 and a minimum score of 3. A lower number indicating a more severe injury and a poorer prognosis.
Change in Glasgow outcome scale (GOS) score | 12 months
  The Glasgow outcome score (GOS) applies to patients with brain damage allowing the objective assessment of their recovery. This allows a prediction of the long-term course of rehabilitation to return to work and everyday life. Scale consists of five grades from 1 to 5. 1 denotes death. 2 denotes persistent vegetative state.3 denotes severe disability. 4 denotes moderate disability and 5 denotes low disability.
MRI (T1, T2, Flair, DWI) scanning | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided